CLINICAL TRIAL: NCT04847908
Title: Changes in Metabolite Concentrations After a Single High-intensity Interval Exercise Intervention During Treatment for Childhood Cancer - A Pilot Study
Brief Title: The Munich Adrenaline Cancer Study
Acronym: MACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, Sabine Kesting, Dr. rer. medic, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TUM
Record Dates: First submitted 2021-03-31; First posted 2021-04-19 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Childhood Cancer
Keywords: exercise; metabolomics; high-intensity interval exercise intervention
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-intensity interval exercise intervention (Experimental): Change according to definition.
  Interventions: Other: Single high-intensity interval exercise intervention

INTERVENTIONS:
Other: Single high-intensity interval exercise intervention — Study participants perform a single bout of exercise on a cycle ergometer (high-intensity interval exercise intervention) within the first and third cycle of chemotherapy. Following a 2 minute warm-up, the interval protocol comprises 10 intervals à 15 seconds with high intensity and 60 seconds low intensity in-between. Blood samples are taken at t0 pre-exercise (after a 10 minute rest) and at t1 immediately post-exercise via central catheter (Hickman/port).

SUMMARY:
Observational studies report associations between physical activity and survival in some types of adult cancer. In addition, some exercise-induced molecules such as catecholamines (e.g., adrenaline) are known to change cancer cell signalling, proliferation and have been linked to clinical outcomes such as survival. The aim of this study is to analyse changes in adrenaline concentration with a single high-intensity interval exercise intervention on a cycle ergometer in children and adolescents during treatment for cancer and to examine the feasibility of the study concept.

DETAILED DESCRIPTION:
Exercise is generally recommended as an adjunct therapy for adult cancer patients as it counteracts the adverse effects of cancer and its treatment. According to epidemiological data, exercise is also associated with a reduced risk of tumour developement and an improval of survival in some tumours. However, the underlying mechanisms by which exercise affects tumour cells are poorly understood in adult cancer patients and mostly unknown in children. Recent studies demonstrate anti-cancer effects of exercise-induced adrenaline through natural killer cell mobilisation and Hippo signalling. In addition, several exercise-induced molecules such as catecholamines (e.g., adrenaline) are known to change cancer cell signalling, proliferation and have been linked to clinical outcomes such as survival. The aim of this pilot study is the analysation of exercise-induced changes in adrenaline concentration in childhood cancer patients and to show feasibility of the study concept. Following recruitment within the first and third cycle of chemotherapy and consent for study participation, all recruited patients perform a single high-intensity interval exercise intervention on a cycle ergometer. Intensity of the intervals is examined both subjectively via a scale for rate of perceived exertion and objectively via changes in lactate concentration pre- and post-exercise as well as heart rate monitoring. Blood samples are taken by trained personnel staff and prepared for processing (centrifuged, snap-frozen). Changes in adrenaline concentration are measured with a commercial ELISA kit. For further identification of metabolites that change with exercise, a non-biased mass spectrometry metabolomics analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed pediatric cancer or relapse
* aged 6-18 years
* between the first and third cycle of chemotherapy
* diagnosis and treatment at the Kinderklinik München Schwabing, Department of Paediatrics and Children's Cancer Research Centre, Technical University of Munich
* German language
* informed consent as documented by signature

Exclusion Criteria:

* Any medical contraindication with respect to a high-intensity interval exercise intervention (e.g., cardiovascular complications, comorbidities, bleeding risk, pain, infection, nausea, orthopedic impairment of the lower extremities)
* inability to follow the procedures and understand the intervention and assessment of the study, e.g., due to cognitive impairment, language problems, psychological disorders etc.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in adrenaline concentration | Pre-exercise (at rest, t0) and post-exercise (within 3 min, t1)
  Blood samples are collected at rest pre-exercise (t0) and post-exercise (t1) via a central catheter and prepared for processing by trained personnel (centrifuged, snap-frozen). Both at t0 and t1, 4,9ml blood are taken for adrenaline and lactate concentration (see secondary outcomes). Serum adrenaline concentration is measured with an ELISA kit in mmol/l.

SECONDARY OUTCOMES:
Feasibility of the study concept | Through study completion, on average 14 days
  Feasibility of the study concept is examined via compliance, acceptance and safety.
  Detailed documentation ensures completeness of feasibility aspects.
Lactate concentration | Pre-exercise (at rest, t0) and post-exercise (within 3 min, t1)
  Lactate concentration is analysed to examine the level of intensity of the single high-intensity interval exercise intervention. Blood samples are collected at rest pre-exercise (t0) and post-exercise (t1), both 4,9ml, via a central catheter and prepared for processing by trained personnel. Lactate concentration is measured with Biosen C-Line in mmol/l.
Heart rate | Pre-exercise (at rest, t0), during high-intensity interval exercise intervention and post-exercise (within 3 min, t1)
  Heart rate monitoring is used to objectively measure the level of intensity during the single high-intensity interval exercise intervention for safety monitoring. Heart rate levels are documented at rest pre-exercise, after every interval and post-exercise.
Physical activity before diagnosis | Once, pre-intervention
  Physical activity levels are investigated using a standardised questionnaire (ActiOn) to evaluate the extent, range and intensity of physical activity shortly before the diagnosis. This questionnaire was developed for children and adolescents during and after treatment for childhood cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Teichert-von Lüttichau, PD Dr. med., Principal Investigator — TUM
Locations (1):
- Kinderklinik München Schwabing, TUM School of Medicine, Department of Paediatrics and Children's Cancer Research Center, Technical University of Munich, Germany, Munich, Germany